CLINICAL TRIAL: NCT05603442
Title: Thoracic Intervertebral Foramen Block: a Prospective Cadaveric Study
Brief Title: Thoracic Intervertebral Foramen Block
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: San Salvatore Hospital of L'Aquila (Other)
Responsible Party: Principal Investigator, Emiliano Petrucci, Medical doctor, San Salvatore Hospital of L'Aquila
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 133/22
Record Dates: First submitted 2022-10-21; First posted 2022-11-02 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Anesthesia; Functional; Anesthesia, Local; Spinal Cord

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thoracic intervertebral foramen block (Experimental): The thoracic intervertebral foramen block is performed at second (T2), fifth (T5), ninth (T9), and twelfth (T12) thoracic vertebra. The ultrasonography is performed by using a high-frequency linear-array ultrasound transducer. A Tuohy needle is inserted in-plane to the ultrasound beam in a lateral-to-medial direction gently to contact the spinous process, into the skeletal muscle plane of the erector spinae muscle. Then, the needle tip is moved to reach the angle between the transverse process and spinous process. Subsequently, the needle tip is gently inserted and advanced for 2 mm along with the superior limit of the vertebral pedicle, until losing contact with the bone. Five ml methylene blue 1% dye (MB) are subsequently injected. The anesthetic procedure is bilaterally performed. Two continuous catheter sets were used and threaded 1 cm from the needle tip, for a bilateral continuous block. The catheters are inserted from the caudal to the cephalic direction.
  Interventions: Procedure: Thoracic intervertebral foramen block

INTERVENTIONS:
Procedure: Thoracic intervertebral foramen block — The thoracic intervertebral foramen block is performed by placing the needle tip over and behind the transverse process of vertebra, via the thoracic intervertebral foramen.

SUMMARY:
The investigators hypothesize an alternative way to perform thoracic paravertebral block, by placing the needle tip over and behind the transverse process of vertebra, via the thoracic intervertebral foramen. This anesthetic procedure is called thoracic intervertebral foramen block.

The study aims to verify the spread of dye on to the the nervous structures of retropleural space (the ventral rami, the communicating rami, and the sympathetic trunk), and into the thoracic paravertebral space and epidural space. To accomplish this, a prospective cadaveric study was designed.

DETAILED DESCRIPTION:
This is a prospective cadaveric study. The anesthetic procedure is performed on 2 corpses for which autopsy is requested, in accordance with Italian Low.

Before performing the autopsy, the corps is placed in the left and then in the right lateral position, to perform bilateral block. The anesthetic procedure is performed at second (T2), fifth (T5), ninth (T9), and twelfth (T12) thoracic vertebra. The ultrasonography is performed by using a high-frequency linear-array US transducer. A Tuohy needle is inserted in-plane to the ultrasound beam in a lateral-to-medial direction gently to contact the spinous process, into the skeletal muscle plane of the erector spinae muscle. Then, the needle tip is moved to reach the angle between the transverse process and spinous process. Subsequently, the needle tip is gently inserted and advanced for 2 mm along with the superior limit of the vertebral pedicle, until losing contact with the bone. Five ml methylene blue 1% dye (MB) were subsequently injected. The anesthetic procedure is bilaterally performed. Two continuous catheter sets are used and threaded 1 cm from the needle tip, for a bilateral continuous block. The catheters are inserted from the caudal to the cephalic direction.

At the end of the anesthetic procedure, a second look ultrasound scan of thoracic paravertebral space was performed. Subsequently, the corps is put in supine position, and autopsy is started.

ELIGIBILITY:
Inclusion Criteria:

* corps for which autopsy is required

Exclusion Criteria:

* corps under Legal custody of Italian Low

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Retropleural spread | During autopsy
  Assess mL of dye on to the nervous structures of retropleural space (the ventral rami, the communicating rami, and the sympathetic trunk)
Thoracic paravertebral spread | During autopsy
  Assess mL of dye on to the thoracic paravertebral space
Epidural spread | During autopsy
  Assess mL of dye on the epidural space

SECONDARY OUTCOMES:
Iatrogenic damages | During autopsy
  Number of punctures of vertebral blood vessels, spinal nerve roots, and pleura
Distance (mm) between the catheter tip and the thoracic intervertebral foramen content is also evaluated | During autopsy
  Distance (mm) between the catheter tip and the thoracic intervertebral foramen content is evaluated
Second look ultrasound scan | After the anesthetic procedure
  Area (square cm) of anechoic shadow on the paravertebral space

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Petrucci, MD, Principal Investigator — San Salvatore Acadeci Hospital of L'Aquila (Italy)
Locations (1):
- San Salvatore Academic Hospital of L'Aquila, L’Aquila, L'Aquila, Italy

IPD SHARING:
Plan to Share IPD: No